CLINICAL TRIAL: NCT06987474
Title: Capella Scientia (SCDX) Development Study
Brief Title: Capella Scientia Development Study
Status: Recruiting | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CTK378-E006
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Subjects/eyes previously implanted with an Alcon monofocal or multifocal presbyopia correcting IOL. Measurements will be taken with Unity DX and SMARTCataract DX (SCDX) Biometer and either the IOLMaster 700 Biometer or the Argos with Alcon Image Guidance Biometer depending on which device is used at site.
  Interventions: Device: Unity DX and SMARTCataract DX (SCDX) Biometer; Device: IOLMaster 700 Biometer; Device: Argos with Alcon Image Guidance Biometer
- Group 2: Subjects/eyes with planned implantation of an Alcon monofocal or monofocal toric IOL. Measurements will be taken with Unity DX and SMARTCataract DX (SCDX) Biometer and either the IOLMaster 700 Biometer or the Argos with Alcon Image Guidance Biometer depending on which device is used at site.
  Interventions: Device: Unity DX and SMARTCataract DX (SCDX) Biometer; Device: IOLMaster 700 Biometer; Device: Argos with Alcon Image Guidance Biometer
- Group 3: Subjects/eyes with with prior refractive surgery such as LASIK or PRK and planned implantation of an Alcon monofocal or monofocal toric IOL. Measurements will be taken with Unity DX and SMARTCataract DX (SCDX) Biometer and either the IOLMaster 700 Biometer or the Argos with Alcon Image Guidance Biometer depending on which device is used at site.
  Interventions: Device: Unity DX and SMARTCataract DX (SCDX) Biometer; Device: IOLMaster 700 Biometer; Device: Argos with Alcon Image Guidance Biometer
- Group 4: Subjects/eyes with keratoconus, a progressive cornea disorder. Measurements will be taken with Unity DX and SMARTCataract DX (SCDX) Biometer and either the IOLMaster 700 Biometer or the Argos with Alcon Image Guidance Biometer depending on which device is used at site.
  Interventions: Device: Unity DX and SMARTCataract DX (SCDX) Biometer; Device: IOLMaster 700 Biometer; Device: Argos with Alcon Image Guidance Biometer

INTERVENTIONS:
Device: Unity DX and SMARTCataract DX (SCDX) Biometer — Unity DX is a CE-marked, noninvasive, noncontact instrument that generates a 3D model of the eye using hyper parallel optical coherence tomography (HP OCT), aberrometry, and topography. The current version of SCDX software will be used in this study.
Device: IOLMaster 700 Biometer — The IOLMaster 700 Biometer is a CE-marked, noninvasive, noncontact instrument that captures optical biometry. Data will be collected using standard clinical assessments.
Device: Argos with Alcon Image Guidance Biometer — The Argos with Alcon Image Guidance biometer is a CE-marked, noninvasive, noncontact instrument that will capture optical biometry. Data will be collected using standard clinical assessments.

SUMMARY:
This study involves collecting biometry and aberration data using the next generation biometer, Unity DX.

DETAILED DESCRIPTION:
In this prospective, noninterventional, single-arm, unmasked, multicenter study, 4 different subject cohorts will be enrolled simultaneously to collect biometry and aberrometry data using Unity DX. This study will be conducted in India, Spain, and the Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an IRB/IEC approved consent form;
* Willing and able to attend study visit(s) as required by the protocol;
* Consenting age at the jurisdiction of study site;
* Other group-specific, protocol required inclusion criteria may apply.

Exclusion Criteria:

* Women of child-bearing potential;
* Unable to fixate due to nystagmus or other eye movement abnormality (e.g., significant strabismus);
* Unclear optical media preventing data capture from all devices in the study;
* Contraindicated for pupil dilation (e.g., narrow angles, allergies) per investigator's clinical judgment;
* Any ocular disease and/or condition that, in the investigator's clinical judgment, may put the subject at significant risk, may compromise study results, or may interfere significantly with the subject's participation in the study;
* Other group-specific, protocol required exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from clinical sites located in India, Spain, and the Philippines.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Manifest Refraction Spherical Equivalent (MRSE) | Group 1 and Group 4: Day 0; Group 2 and Group 3: Screening (Day -30 to Day -1), Day 30 to 60 postoperative, Day 70 to 100 postoperative
  A manifest refraction (manual refraction) will be performed using a phoropter. The spherical equivalent is calculated by adding the sum of the sphere power with half of the cylinder power. MRSE will be reported in diopters.

CONTACTS AND LOCATIONS:
Overall Officials: Principal II, Clinical Trial Operations, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- Narayana Nethralaya, Bangalore, India
- Asian Eye Institute, Makati City, Philippines
- Spain (2):
  - Clinica Novovision - Clinica Madrid, Madrid
  - Clinica Rementeria, Madrid

IPD SHARING:
Plan to Share IPD: No